CLINICAL TRIAL: NCT03506152
Title: Prospective Evaluation of Serum Procalcitonin in Critically Ill Patients With Suspected Sepsis- Experience From a Tertiary Care Hospital in Pakistan
Brief Title: Evaluation of Serum Procalcitonin in Critically Ill Patients With Suspected Sepsis
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sibtain Ahmed, Consultant, Aga Khan University
Other Study IDs: RRG # 2013-06
Record Dates: First submitted 2018-04-12; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Culture positive
  Interventions: Diagnostic Test: Serum Procalcitonin
- Culture negative
  Interventions: Diagnostic Test: Serum Procalcitonin

INTERVENTIONS:
Diagnostic Test: Serum Procalcitonin — Seven ml of blood was drawn in gel separator tubes within 24 hours of admission in ICU for Procalcitonin determination

SUMMARY:
Procalcitonin is a promising marker of sepsis in critically ill patients. Procalcitonin have better diagnostic accuracy compared to White blood cell count and C - reactive protein. Investigators propose that adding Procalcitonin to the list of standard laboratory work up of critically ill patients with suspected sepsis could increase diagnostic accuracy leading to better patient care.

DETAILED DESCRIPTION:
Background: Sepsis is the leading cause of mortality in critically ill patients. Procalcitonin (PCT) is a promising marker for identification of bacterial sepsis. The aim of this study was to determine the diagnostic accuracy of serum PCT concentration in patients with suspected sepsis admitted to mixed medical-surgical Intensive care unit (ICU).

Material and Methods: A cross-sectional study conducted at section of Chemical Pathology, Department of Pathology and Laboratory Medicine and ICU. Patients with suspected sepsis were included, serum PCT cut off ≥0.5 ng /ml was taken for diagnosing sepsis. Diagnostic accuracy was measured in terms of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) taking blood culture as gold standard. Furthermore, different cut offs were compared by using receiver operating characteristic curves (ROC). Data analysis was done on SPSS version.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients less than 70 and greater than 18 years of age
2. Patients full filling the sepsis definition (American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference)
3. Patients were recruited within 24 hour of ICU admission

Exclusion Criteria:

1. Patients discharged before 24 hours
2. Patients who had blood transfusion before ICU stay
3. Patients with organ failure

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with suspected sepsis were recruited
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2015-12-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of Procalcitonin | one year
  Diagnostic accuracy was measured in terms of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) taking blood culture as gold standard. Furthermore, different cut offs were compared by using receiver operating characteristic curves (ROC).

CONTACTS AND LOCATIONS:
Locations (1):
- Sibtain Ahmed, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No